CLINICAL TRIAL: NCT06012916
Title: Brain Network Dynamics of Depression During Esketamine Treatment
Acronym: K-BRAINED
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0696
Record Dates: First submitted 2023-07-14; First posted 2023-08-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depressive Disorder, Major
Keywords: Esketamine; Ketamine; Belief Updating; Pupillometry; EEG
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Esketamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment Resistant Depression + Esketamine Treatment: This is a group of individuals with treatment resistant depression receiving Esketamine treatment as prescribed by their physician during outpatient appointments over several weeks at the Interventional Psychiatry outpatient clinic at University of North Carolina at Chapel Hill (UNC). After signing the informed consent, electroencephalogram (EEG) will be recorded before and after Esketamine administration by the attending physician. The participant will perform a cognitive task before and after the Esketamine administration as well as complete self-scored questionnaire regarding depressive symptoms, treatment expectation and Esketamine side-effects. Clinical information like the duration of episode, medication or clinician-rated depression scores will be retrieved from the charting system.
  Interventions: Drug: Esketamine nasal spray

INTERVENTIONS:
Drug: Esketamine nasal spray — This is an observational study. The Esketamine nasal spray is administered by the attending physician during a regular treatment appointment at the Interventional Psychiatry Clinic. Esketamine dosages may range between 28-84mg. The study does not interfere with the individual treatment plan in any way.
  Other Names: Spravato

SUMMARY:
This is a monocentric, observational clinical trial investigating the effect of Esketamine on brain network activity and a belief updating task in people with depression. We investigate the immediate and the long-term effect (approx. 8 weeks) of Esketamine on EEG signals, pupillometry and belief updating and the relation of those effects on depressive symptomatology.

DETAILED DESCRIPTION:
The FDA approved the S-enantiomer of Ketamine in a nasal spray formulation (Esketamine, Spravato) in 2019 for treatment resistant depression in conjunction with an oral antidepressant. Albeit showing impressive short term clinical effects, the neurophysiological mechanism leading to clinical improvements are not understood. The investigators aim to add missing knowledge about the network dynamics of Esketamine in depression. Besides changes of neural signatures, Esketamine might impact cognitive processes like belief updating.

Previous studies have shown that people update their expectations of future life events after receiving novel information. The Belief Updating Task (BUT) measures this belief update in reaction to new information. Healthy individuals have been shown to update their beliefs "optimistically", making larger changes in their expectations in response to good news. Individuals with depression lack this optimistic belief update bias. Therefore, the investigators also aim to examine if Esketamine treatment reinstates the optimistic bias, how those changes are mediated by neurophysiological changes during the task and if a change in belief updated is related to a change of depressive symptoms.

The first session takes place at the start of the Esketamine treatment period, whereas the second experimental session is conducted closer to the end of the treatment period. In both experimental sessions, EEG/pupillometry and cognitive measurements are taken before and after Esketamine administration. Analyses will assess pre/post Esketamine effects within a session and between two sessions.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder
* Receiving Esketamine nasal spray treatment for depression
* Ability to understand study procedures and sign an informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The goal is to recruit individuals with an MDD diagnosis who are receiving Esketamine treatment.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Belief Updating in Session 1 | 10 minutes before Esketamine application compared to 2 hours after Esketamine application
  Participants rate the likelihood of a negative life event happening to them (E1) and their confidence in the estimate (C1). They are given a base rate (BR), described as the average lifetime probability of that event happening to someone with the same demographics. Participants will then again rate how likely the event could happen to them personally (E2).
  Outcome variables: update = |E2 - E1| and estimation error (ER) = |E1 - BR| News: "good news" (BR< E1) or "bad news" (BR>E1) trials.
  Within session relationships between update, C1, ER and covariates will be investigated using linear mixed models (LMMs) using an iterative model comparison process. The basic model will include fixed effect of News and a random intercept for individuals (id or ID).
  Potential covariates likely include ER, C1, the Revised Life Orientation Test (LOT-R), Ketamine Side Effect Tool (KSET), and scores of depression severity.
Change in Belief Updating in Session 2 | 10 minutes before Esketamine application compared to 2 hours after Esketamine application
  Participants rate the likelihood of a negative life event happening to them (E1) and their confidence in the estimate (C1). They are given a base rate (BR), described as the average lifetime probability of that event happening to someone with the same demographics. Participants will then again rate how likely the event could happen to them personally (E2).
  Outcome variables: update = |E2 - E1| and estimation error (ER) = |E1 - BR| News: "good news" (BR< E1) or "bad news" (BR>E1) trials.
  Within session relationships between update, C1, ER and covariates will be investigated using linear mixed models (LMMs) using an iterative model comparison process. The basic model will include fixed effect of News and a random intercept for ID (individuals).
  Potential covariates likely include ER, C1, the Revised Life Orientation Test (LOT-R), Ketamine Side Effect Tool (KSET), and scores of depression severity.
Change in Confidence in Beliefs Questionnaire in Session 1 | 30 minutes before Esketamine application compared to 2 hours after Esketamine application
  * Confidence in Beliefs Questionnaire investigates the strengths of belief in statements about the participant and about someone close to them.
  * Participants rate how certain they are about each belief, higher values imply higher certainty
  * Beliefs about oneself: 12 items (6 positive, 6 negative), Likert Scale 0 to 100, participants make a mark on a line
  * Beliefs about others: 12 items (6 positive, 6 negative), Likert Scale 0 to 100, participants make a mark on a line
Change in Confidence in Beliefs Questionnaire in Session 2 | 30 minutes before Esketamine application compared to 2 hours after Esketamine application
  * Confidence in Beliefs Questionnaire investigates the strengths of belief in statements about the participant and about someone close to them.
  * Participants rate how certain they are about each belief, higher values imply higher certainty
  * Beliefs about oneself: 12 items (6 positive, 6 negative), Likert Scale 0 to 100, participants make a mark on a line
  * Beliefs about others: 12 items (6 positive, 6 negative), Likert Scale 0 to 100, participants make a mark on a line
Change of Ketamine Side Effect Tool (KSET) in Session 1 | 5 minutes before Esketamine application, and 50, 95, and 130 minutes after Esketamine application
  * Semi-structured interview to assess side effects of ketamine
  * Each item is scores from 0 (=never) to 3 (= severe) points
  * Sum scores and individual item scores can be analyzed.
Change of Ketamine Side Effect Tool (KSET) in Session 2 | 5 minutes before Esketamine application, and 50, 95, and 130 minutes after Esketamine application
  * Semi-structured interview to assess side effects of ketamine
  * Each item is scores from 0 (=never) to 3 (= severe) points
  * Sum scores and individual item scores can be analyzed.
Change in Mood Likert Scale in Session 1 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes after Esketamine application
  * Likert Scales range from 0 to 100
  * Participants make a mark on a line (left end = 0, right end = 100)
Change in Mood Likert Scale in Session 2 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes after Esketamine application
  * Likert Scales range from 0 to 100
  * Participants make a mark on a line (left end = 0, right end = 100)
Change in Quality of Life Enjoyment and Satisfaction Questionnaire, short version (Q-LES-Q-SF) | Session 1 and session 2
  * Change in Q-LES-Q-SF between Session 1 and Session 2
  * Q-LES-Q-SF is a brief, self-scoring quality of life rating scale.
  * Maximum percentage is 100%. Higher values imply higher quality of life
Change in Patient Health Questionnaire (PHQ-9) | Session 1 and session 2
  * Change in PHQ-9 between Session 1 and Session 2
  * PHQ-9 is a brief, self-scoring depression rating scale. Higher values imply a higher depression severity.
  * Cut-off for depression is considered >4 PHQ-9 points
Change in Hamilton Depression Rating Scale (HDRS) | Session 1 and session 2
  * Change in HDRS-17 between Session 1 and Session 2
  * HDRS-17 is the most established depression rating scale. Higher values imply a higher depression severity.
  * Cut-off for depression is considered >8 HDRS-17 points
Change of Resting State EEG - Power in Session 1 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and130 minutes after Esketamine application
  * Changes in oscillatory power within an experimental session pre/post Esketamine application
  * Power will be analyzed in canonical frequency bands (e.g. alpha, beta, gamma, delta, theta)
Change of Resting State EEG - Power in Session 2 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and130 minutes after Esketamine application
  * Changes in oscillatory power within an experimental session pre/post Esketamine application
  * Power will be analyzed in canonical frequency bands (e.g. alpha, beta, gamma, delta, theta)
Change of Resting State EEG - Connectivity in Session 1 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes after Esketamine application
  - Changes in functional connectivity in canonical frequency band within an experimental session pre/post Esketamine application
Change of Resting State EEG - Connectivity in Session 2 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes after Esketamine application
  - Changes in functional connectivity in canonical frequency band within an experimental session pre/post Esketamine application
Change of Resting State EEG - Source in Session 1 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes after Esketamine application
  - Changes in spatial distribution and source of electric activity in canonical frequency band within an experimental session pre/post Esketamine application
Change of Resting State EEG - Source in Session 2 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes after Esketamine application
  - Changes in spatial distribution and source of electric activity in canonical frequency band within an experimental session pre/post Esketamine application
Change of Resting State EEG - Aperiodic Signal in Session 1 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes after Esketamine application
  - Changes in slope and offset of the aperiodic EEG signal within an experimental session pre/post Esketamine application
Change of Resting State EEG - Aperiodic Signal in Session 2 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes after Esketamine application
  - Changes in slope and offset of the aperiodic EEG signal within an experimental session pre/post Esketamine application
Change of Resting State EEG - Entropy in Session 1 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes in after Esketamine application
  - Changes of entropy measured in Lempel-Ziv Complexity and mutual information within an experimental session pre/post Esketamine application
Change of Resting State EEG - Entropy in Session 2 | 5 minutes before Esketamine application, and 15, 35, 50, 75, 95, and 130 minutes after Esketamine application
  - Changes of entropy measured in Lempel-Ziv Complexity and mutual information within an experimental session pre/post Esketamine application

SECONDARY OUTCOMES:
Change in Task EEG - Event Related Potential (ERP) in Session 1 | 30 minutes before Esketamine application and 100 minutes after Esketamine application
  * ERP after presentation of baseline will be calculated for trials with good/bad news, low/high estimation error and low/high confidence (-500 to 2000ms)
  * We will analyze the amplitude and spatial distribution of canonical ERP such as N1,N2, P3 and late positive potential
Change in Task EEG - Event Related Potential (ERP) in Session 2 | 30 minutes before Esketamine application and 100 minutes after Esketamine application
  * ERP after presentation of baseline will be calculated for trials with good/bad news, low/high estimation error and low/high confidence (-500 to 2000ms)
  * We will analyze the amplitude and spatial distribution of canonical ERP such as N1,N2, P3 and late positive potential
Change in Task EEG - Time Frequency Analysis in Session 1 | 30 minutes before Esketamine application and 100 minutes after Esketamine application
  * Using wavelet convolution we will conduct a time-frequency analysis for good/bad news, low/high estimation error and low/high confidence
  * Time of interest -500 to 2000ms after base rate presentation
  * Frequency of interest will be 2-40Hz
Change in Task EEG - Time Frequency Analysis in Session 2 | 30 minutes before Esketamine application and 100 minutes after Esketamine application
  * Using wavelet convolution we will conduct a time-frequency analysis for good/bad news, low/high estimation error and low/high confidence
  * Time of interest -500 to 2000ms after base rate presentation
  * Frequency of interest will be 2-40 Hertz (Hz)
Change in Pupillometry in Session 1 | 30 minutes before Esketamine application and 100 minutes after Esketamine application
  * Pupil size during good/bad news and high/low estimation error and low/high confidence trials in the belief updating task
  * Time-locked around the presentation of the base rate (-500 to 2000ms)
Change in Pupillometry in Session 2 | 30 minutes before Esketamine application and 100 minutes after Esketamine application
  * Pupil size during good/bad news and high/low estimation error and low/high confidence trials in the belief updating task
  * Time-locked around the presentation of the base rate (-500 to 2000ms)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Center for Neurostimulation, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No